CLINICAL TRIAL: NCT05948826
Title: A Phase 1, First in Human, Dose-Escalation Study of TORL-3-600 in Participants With Advanced Cancer
Brief Title: First in Human Study of TORL-3-600 in Participants With Advanced Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TORL Biotherapeutics, LLC (Industry)
Collaborators: Translational Research in Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TORL3600-001
Record Dates: First submitted 2023-07-09; First posted 2023-07-17 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumor; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Monotherapy Dose Dose Finding - Part 1 (Experimental): TORL-3-600
  Interventions: Drug: TORL-3-600
- Expansion as Monotherapy - Part 2 (Experimental): TORL-3-600
  Interventions: Drug: TORL-3-600

INTERVENTIONS:
Drug: TORL-3-600 — antibody drug conjugate

SUMMARY:
This first-in-human study will evaluate the safety, tolerability, pharmacokinetics, and antitumor activity of TORL-3-600 in patients with advanced cancer

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumor
* Measurable disease, per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate organ function

Exclusion Criteria:

* Has not recovered [recovery is defined as NCI CTCAE, version 5.0, grade ≤1] from the acute toxicities of previous therapy, except treatment-related alopecia or laboratory abnormalities otherwise meeting eligibility requirements
* Received prior chemotherapeutic, investigational, or other therapies for the treatment of cancer within 14 days with small molecule and within 28 days with biologic before the first dose of TORL-3-600
* Progressive or symptomatic brain metastases
* Serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection
* History of significant cardiac disease
* History of myelodysplastic syndrome (MDS) or AML
* History of another cancer within 3 years before Day 1 of study treatment, with the exception of basal or squamous cell carcinoma of the skin that has been definitively treated. A history of other malignancies with a low risk of recurrence, including appropriately treated ductal carcinoma in situ (DCIS) of the breast and prostate cancer with a Gleason score less than or equal to 6, are also not excluded
* If female, is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2026-06-25 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events and serious adverse events | up to 2 years
  Incidence and severity of adverse events, serious adverse events, according to NCI-CTCAE Version 5.0
Maximum Tolerated Dose (MTD) | 28 Days
  Highest administered dose with < 33% participants experiencing dose limiting toxicity (DLT) in the first 6 DLT evaluable participants
Recommended Phase 2 Dose (RP2D) | up to 2 years
  Based on the maximum tolerated dose, cumulative safety, and pharmacokinetic data

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 2 years
  Percentage of participants with best response of complete response (CR) or partial response (PR) according to RECIST 1.1
Duration of Response (DOR) | up to 2 years
  Time from CR or PR to objective disease progression or death to any cause
Progression Free Survival (PFS) | up to 2 years
  PFS is defined as the time from the start of the treatment until objective disease progression or death from any cause
Time to Response (TTR) | up to 2 years
  Time from start of treatment to complete response or partial response
1 Year Overall Survival (1YOS) | 1 year
  Proportion of participants alive at 1 year from the start of treatment to death from any cause
2 Year Overall Survival (2YOS) | 2 years
  Proportion of participants alive at 2 years from the start of treatment to death from any cause
Number of anti-drug antibody (ADA) Positive Participants | up to 2 years
  Immunogenicity will be measured by the number of participants that are ADA positive.
Maximum Serum Concentration of TORL-3-600 (Cmax) | 21 days
  PK assessment
Minimum Serum Concentration of TORL-3-600 (Cmin) | 21 days
  PK assessment
Maximum Serum Concentration of TORL-3-600 at Steady State (Cmax,ss) | 63 days
  PK assessment
Minimum Serum Concentration of TORL-3-600 at Steady State (Cmin,ss) | 63 days
  PK assessment
Time of Maximum Serum Concentration of TORL-3-600 (Tmax) | 21 days
  PK assessment
Time of Minimum Serum Concentration of TORL-3-600 (Tmin) | 21 days
  PK Assessment
Time of Minimum Serum Concentration of TORL-3-600 at Steady State (Tmin,ss) | 63 days
  PK Assessment
Terminal Half-life (t1/2) of Serum TORL-3-600-ADC | 63 days
  PK Assessment
Area under the Serum Concentration-Time curve from the time of dosing to the last measurable concentration (AUClast) for TORL-3-600 | 21 days
  PK Assessment
Area under the Serum Concentration-Time curve from the time of dosing extrapolated to time infinity (AUCinf) for TORL-3-600 | 63 days
  PK Assessment
Apparent volume of distribution during the terminal phase (Vz) of TORL-3-600 | 63 days
  PK Assessment
Clearance (CL) of TORL-3-600 | 63 days
  PK Assessment
Accumulation ratio (Rac) of TORL-3-600 | 63 days
  PK Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Labib, PharmD, Study Chair — TORL Biotherapeutics, LLC
Locations (9):
- United States (7):
  - Providence Medical Foundation, Fullerton, California
  - UCLA - JCCC Clinical Research Unit, Los Angeles, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - Fort Wayne Medical Oncology and Hematology Inc., Fort Wayne, Indiana
  - Washington University School of Medicine-Siteman Cancer Center, St Louis, Missouri
  - Sarah Cannon Research Institute-Tennessee, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
- Canada (2):
  - University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No